CLINICAL TRIAL: NCT06709339
Title: A Phase IV, Multicentre, Open-label, Single-arm Study to Investigate the Efficacy, Safety and Durability of Faricimab (RO6867461) in Caucasian Patients With Polypoidal Choroidal Vasculopathy
Brief Title: Study to Investigate the Efficacy, Safety and Durability of Faricimab in Caucasian Patients With Polypoidal Choroidal Vasculopathy (MONDEGO)
Acronym: MONDEGO
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Association for Innovation and Biomedical Research on Light and Image (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ECR-AMD-2024-15; 2024-515640-22-00 (EU CTIS Number)
Record Dates: First submitted 2024-11-25; First posted 2024-11-29 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Polypoidal Choroidal Vasculopathy
Keywords: Faricimab; Caucasian patients; PCV; Durability; Safety; Efficacy
MeSH Terms: conditions — Polypoidal Choroidal Vasculopathy | interventions — faricimab

STUDY DESIGN:
Intervention Model Description: This study will be conducted in adult Caucasian participants with symptomatic macular PCV, a subtype of nAMD, which was under-represented in the faricimab Phase III pivotal Studies TENAYA (ClinicalTrials.gov identifier: NCT03823287) and LUCERNE (ClinicalTrials.gov identifier: NCT03823300) where less than 2% of the enrolled participants with nAMD were diagnosed with PCV and no Caucasian participants with symptomatic macular PCV were identified in the mentioned pivotal Studies.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Faricimab (Experimental): This open-label, single-arm study will evaluate the efficacy, safety, and durability of Faricimab Injection [Vabysmo] 6 mg anti-VEGF IVT in Caucasian patients with symptomatic macular PCV.
  Interventions: Drug: Faricimab Injection [Vabysmo]

INTERVENTIONS:
Drug: Faricimab Injection [Vabysmo] — The investigational medicinal product (IMP) for this study is faricimab (RO6867461), as per clinical practice. No control treatment will be used for this study

SUMMARY:
The goal of this clinical trial is to assess the efficacy, safety and durability of faricimab in caucasian patients with polypoidal choroidal vasculopathy (PCV). The main question it aims to answer is:

To evaluate the efficacy of intravitreal (IVT) injections of faricimab 6 milligrams (mg) on Best Corrected Visual Acuity (BCVA) outcomes in caucasian patients with symptomatic macular PCV.

Participants will undergo ophthalmic examination, safety assessment and treatment with faricimab according to a patient specific treat and extend regimen.

DETAILED DESCRIPTION:
Polypoidal choroidal vasculopathy (PCV) was first described in 1982 by Yannuzzi as a choroidal vasculopathy leading to haemorrhagic and exudative macular degeneration. More than four decades later, the pathogenesis of the disease remains uncertain with authors considering PCV a subtype of neovascular age-related macular degeneration (nAMD) while others advocate a separate clinical entity and adequate treatment is still an unmet need.

Several studies have reported an association between PCV and major and minor interethnic classification differences regarding morphological alterations, prevalence, genetic associations, lesion location, and results after anti-vascular endothelial growth factor (VEGF) treatment, among others. For instance, the reported prevalence of PCV in patients with neovascular AMD ranges from 4% to 9,8% in Caucasians and from 22% to 55% in Asians. However, a recent study reported a much higher prevalence in Caucasians (22,1%), suggesting that PCV may actually be underdiagnosed in this population.

Today, intravitreal (IVT) anti-VEGF therapy plays a key role in the management of PCV and has become the standard of care. The anti-permeability property of anti-VEGF agents, such as aflibercept and ranibizumab, play a role in reducing the exudation from abnormal choroidal vessels and polypoidal lesions, thereby decreasing the subretinal fluid and preserving vision.

Although the current standard of care has demonstrated clinical benefit for patients with PCV, many limitations exist in understanding the disease as a result of its heterogeneity in clinical features and treatment outcomes. The burden of frequent injections, incomplete polypoidal lesion closure, and the risk and unpredictability of lesion relapse reinforce the need to develop new treatments for patients with PCV. This population is at risk of disease relapse, retinal haemorrhage, and vision loss, and is appropriate for inclusion in this clinical trial.

Faricimab is a novel humanized bispecific Immunoglobulin G1 (IgG1) monoclonal antibody that selectively binds with high affinity to VEGF-A and angiopoietin-2 (Ang-2). Faricimab was studied for the treatment of neovascular AMD (nAMD) in the global Phase III Studies TENAYA (ClinicalTrials.gov identifier: NCT03823287) and LUCERNE (ClinicalTrials.gov identifier: NCT03823300) and is currently being studied in the long-term extension Study AVONELLE-X (ClinicalTrials.gov identifier: NCT04777201). The TENAYA (ClinicalTrials.gov identifier: NCT03823287) and LUCERNE (ClinicalTrials.gov identifier: NCT03823300) studies consistently showed that faricimab, given at intervals of up to 16 weeks, offered non-inferior vision gains compared with aflibercept, given every 2 months in the first year. Approximately 50% of participants eligible for extended dosing with faricimab were able to be treated every 4 months, and nearly 80% of participants every 3 months or longer. However, patients with symptomatic macular PCV were under-represented in the faricimab Phase III pivotal Studies TENAYA (ClinicalTrials.gov identifier: NCT03823287) and LUCERNE (ClinicalTrials.gov identifier: NCT03823300).

The purpose of this study is to assess the efficacy, durability, and safety of faricimab 6 mg IVT administered at up to 24-week intervals in the treatment-naive study eye of Caucasian patients with symptomatic macular PCV. This study will add to the evidence base for the benefit-risk profile of faricimab IVT injection in Caucasian patients with symptomatic macular PCV.

The study consists of a screening period of up to 28 days (Days -28 to -1) in length and an approximately 100-week study treatment period consisting of a Treatment Initiation period (Weeks 1-12) and the treat and extend (T&E) regimen period (Weeks 20-Week 100).

ELIGIBILITY:
General Inclusion Criteria:

Potential participants are eligible to be included in the study only if all of the following criteria apply:

* Signed ICF
* Age ≥ 50 years at the time of signing the ICF
* Caucasian
* Participants who are able to comply with the study protocol, in the investigator's judgment
* For female participants of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraception as defined below:

Female participants must remain abstinent or use contraceptive methods with a failure rate of < 1% per year, during the treatment period and for at least 3 months after the final dose of faricimab.

A female participant is considered to be of childbearing potential if she is post-menarche, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and is not permanently infertile due to surgery (i.e., removal of ovaries, fallopian tubes, and/or uterus) or another cause as determined by the investigator (e.g., Müllerian agenesis). Per this definition, a female participant with a tubal ligation is considered to be of childbearing potential. The definition of childbearing potential may be adapted for alignment with local guidelines or regulations.

Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.

The reliability of sexual abstinence should be evaluated concerning the duration of the clinical trial and the preferred and usual lifestyle of the individual.

Periodic abstinence (e.g., calendar, ovulation, symptothermal, or post-ovulation methods) and withdrawal are not adequate methods of contraception.

If required per local guidelines or regulations, locally recognized adequate methods of contraception and information about the reliability of abstinence will be described in the local ICF.

Ocular Inclusion Criteria for study eye:

* Sufficiently clear ocular media and adequate pupillary dilatation to allow acquisition of good quality retinal images to confirm diagnosis
* Confirmed diagnosis, by the Reading Centre, of naïve symptomatic macular PCV defined by the following:

  * Active macular polypoidal lesions shown by ICGA AND
  * Presence of exudative or haemorrhagic features involving the macula as identified by the investigator using multimodal images.
* BCVA scores of 78-24 ETDRS letters, inclusive (20/32 to 20/320 approximate Snellen equivalent), using the ETDRS protocol and assessed at the initial testing distance of 4 meters [see the BCVA Standard Operational Procedures (SOP) for additional details] on study Day 1.

General Exclusion Criteria

Potential participants are excluded from the study if any of the following criteria apply:

* Treatment with investigational therapy (device, drug, or traditional medicine with the exception of vitamins and minerals) within 3 months prior to initiation of study treatment on study Day 1
* Any major illness or major surgical procedure within 1 month before screening
* Active cancer within the 12 months prior to study Day 1 except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, and prostate cancer with a Gleason score of ≤ 6 (Grade Group of 1) and a stable prostate-specific antigen for ≥ 12 months
* Continuous use of any medications and treatments indicated below:

  * Systemic anti-VEGF therapy
  * Systemic drugs known to cause macular oedema (fingolimod, tamoxifen)
  * Other experimental therapies (except those comprising vitamins and minerals) and therapies that claim to have an effect on macular pathology (e.g., kallidinogenase)
* Systemic treatment for suspected or active systemic infection on study Day 1
* Ongoing use of prophylactic antibiotic therapy may be acceptable after discussion with the Medical Monitor.
* Uncontrolled blood pressure, defined as systolic blood pressure > 180 mmHg and/or diastolic blood pressure > 100 mmHg while the participant is at rest on study Day 1
* History of stroke (cerebral vascular accident) or myocardial infarction within 6 months prior to study Day 1
* History of other diseases, metabolic dysfunction, physical examination finding, or historical or current clinical laboratory findings giving reasonable suspicion of a condition that contraindicates the use of the IMP or that might affect the interpretation of the results of the study or renders the participant at high risk for treatment complications in the opinion of the investigator
* History of severe allergic reaction or anaphylactic reaction to a biologic agent or known hypersensitivity to any component of the faricimab injection, study-related procedure preparations (including fluorescein and indocyanine green dyes), dilating drops, or any of the anaesthetic and antimicrobial preparations used by a participant during the study
* Pregnancy or breastfeeding, or intention of becoming pregnant during the study or within 28 days after the final dose of faricimab

Ocular Exclusion Criteria

Potential participants are excluded from the study if any of the following criteria apply to both eyes:

* History of idiopathic or autoimmune-associated uveitis in either eye
* Active ocular inflammation or suspected or active ocular or periocular infection in either eye on study Day 1

Participants who meet any of the following ocular criteria for the study eye will be excluded from study entry:

* Any history or presence of macular pathology unrelated to PCV affecting vision or contributing to the presence of macular haemorrhage, IRF, or SRF
* Retinal pigment epithelial tear involving the macula on study Day 1
* Diagnosis with or suspected of having narrow-angle glaucoma who have not undergone iridotomy. The inclusion of these patients will be conditional upon prior referral to the relevant specialist for appropriate treatment to enable participation in the study.
* On FFA/colour fundus photograph (CFP):

  * Subretinal haemorrhage of > 4 macular photocoagulation study disc area and/or that involves the fovea
  * Fibrosis or atrophy of > 50% of the total lesion area and/or that involves the fovea
  * Any concurrent intraocular condition (e.g., amblyopia, aphakia, retinal detachment, cataract, diabetic retinopathy or maculopathy, or epiretinal membrane with traction) that, in the opinion of the investigator, could either reduce the potential for visual improvement or require medical or surgical intervention during the study
  * Current vitreous haemorrhage on study Day 1
  * Advanced/or uncontrolled glaucoma
  * Spherical equivalent of refractive error demonstrating more than 8 dioptres of myopia
* Any prior or concomitant treatment for PCV or other retinal diseases, including, but not restricted to, IVT treatment (e.g., faricimab, anti-VEGF, steroids, tissue plasminogen activator, ocriplasmin, C3F8, air), periocular pharmacological intervention, argon laser photocoagulation, verteporfin PDT, diode laser, transpupillary thermotherapy, or ocular surgical intervention
* Any cataract surgery or treatment for complications of cataract surgery with steroids or yttrium-aluminum-garnet (YAG) laser capsulotomy within 3 months prior to study Day 1
* Any other intraocular surgery (e.g., pars plana vitrectomy, glaucoma surgery, corneal transplant, or radiotherapy)
* Prior periocular pharmacological or IVT treatment (including anti-VEGF medication) for other retinal diseases
* Continuous use of any medications and treatments indicated below:

  * IVT anti-VEGF agents (other than study-assigned faricimab)
  * IVT, periocular (subtenon), steroid implants (i.e., Ozurdex®, Illuvien®), or chronic topical ocular corticosteroids (defined as continuous usage for 100 days or longer)
  * Concurrent use of any macular photocoagulation or PDT with verteporfin Participants who have a non-functioning fellow (non-study) eye, defined as either BCVA of hand motion or worse, or no physical presence of non-study eye (i.e., monocular), at both the screening and study Day 1 visits will be excluded from study entry.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-08-06 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in BCVA in the study eye to Week 40 or 44 or 48 | From Baseline through Week 40 or 44 or 48
  Best Corrected Visual Acuity (BCVA) is measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA from baseline indicates an improvement in visual acuity.

SECONDARY OUTCOMES:
Change from Baseline in BCVA in the Study | From baseline through last treatment visit (up to 100 weeks)
  Best Corrected Visual Acuity (BCVA) is measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart
Change from Baseline in BCVA in the Study Eye to the last treatment visit | From Baseline through last treatment visit (up to 100 weeks)
  At a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA from baseline indicates an improvement in visual acuity.
Change From Baseline in BCVA in the Study Eye Over Time | Over time (up to 104 weeks)
  Best Corrected Visual Acuity (BCVA) is measured on the ETDRS chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA from baseline indicates an improvement in visual acuity.
Proportion of Participants Gaining Greater Than or Equal to (≥)15, ≥10, or ≥5 Letters from the Baseline BCVA in the Study Eye Averaged Over Time | Over time (up to 104 weeks)
  Best Corrected Visual Acuity (BCVA) is measured on the ETDRS chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA from baseline indicates an improvement in visual acuity.
Proportion of Participants Avoiding a Loss of ≥15, ≥10, or ≥5 Letters from the Baseline BCVA in the Study Eye Over Time | Over time (up to 104 weeks)
  Best Corrected Visual Acuity (BCVA) is measured on the ETDRS chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score) and avoiding a loss in BCVA from baseline indicates no worsening in visual acuity.
Percentage of Participants Maintaining or Achieving BCVA Snellen Equivalent of 20/40 (BCVA =69 Letters) in the Study Eye | Over time (up to 104 weeks)
  Best Corrected Visual Acuity (BCVA) was measured on the ETDRS chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA letter score from baseline indicates an improvement in visual acuity.
Proportion of participants with complete polypoidal lesion regressions at Weeks 40, 44, or 48 | From Baseline through Week 40 or 44 or 48
  Complete polypoidal lesions regressions are measured using Indocyanine Green Angiography (ICGA), as assessed by the central reading center.
Proportion of participants with complete polypoidal lesion regressions at the end of the study | From Baseline through the end of the study (up to 104 weeks)
  Complete polypoidal lesions regressions are measured using Indocyanine Green Angiography (ICGA), as assessed by the central reading center.
Change From Baseline in Central Subfield Thickness in the Study Eye at Weeks 40 or 44, or 48 | From Baseline through Week 40 or 44 or 48
  Central subfield thickness (CST) is defined as the distance between the internal limiting membrane (ILM) and the retinal pigment epithelium (RPE) using optical coherence tomography (OCT), as assessed by the central reading center.
Change from Baseline in Central Subfield Thickness in the Study Eye to the end of the study | From Baseline through the end of the study (up to 104 weeks)
  Central subfield thickness (CST) is defined as the distance between the ILM and the RPE using OCT, as assessed by the central reading center.
Change From Baseline in Central Subfield Thickness in the Study Eye Over Time | Over time (up to 104 weeks)
  Central subfield thickness (CST) is defined as the distance between the ILM and the RPE using OCT, as assessed by the central reading center.
Proportion of Participants With no Intraretinal Fluid and no subretinal fluid in the Study Eye at Week 20 | From Baseline and Week 20
  Intraretinal fluid and subretinal fluid are measured using OCT in the central subfield (center 1 millimetre [mm]).
Proportion of Participants With no Intraretinal Fluid and no subretinal fluid in the Study Eye at Weeks 40 or 44, or 48 | From Baseline and Week 40 or 44 or 48
  Intraretinal fluid and subretinal fluid are measured using OCT in the central subfield (center 1 mm).
Proportion of Participants With no Intraretinal Fluid and no subretinal fluid in the Study Eye at the end of the study | From Baseline and the end of the study (up to 104 weeks)
  Intraretinal fluid and subretinal fluid are measured using OCT in the central subfield (center 1 mm).
Proportion of Participants With no Intraretinal Fluid, no Subretinal Fluid and no sub-RPE fluid in the Study Eye at Week 20 | From Baseline and Week 20
  Intraretinal fluid, subretinal fluid and sub-RPE fluid are measured using OCT in the central subfield (center 1 mm).
Proportion of Participants With no Intraretinal Fluid, no Subretinal Fluid and no sub-RPE fluid in the Study Eye at Weeks 40 or 44, or 48 | From Baseline and Week 40 or 44 or 48
  Intraretinal fluid, subretinal fluid and sub-RPE fluid are measured using OCT in the central subfield (center 1 mm).
Proportion of Participants With no Intraretinal Fluid, no Subretinal Fluid and no sub-RPE fluid in the Study Eye at the end of the study | From Baseline and the end of the study (up to 104 weeks)
  Intraretinal fluid, subretinal fluid and sub-RPE fluid are measured using OCT in the central subfield (center 1 mm).
Change From Baseline in branch Neovascularization network in the Study Eye at 1 year | Baseline and 1 year
  The branch neovascularization network in the study eye is evaluated by a central reading center using OCT angiography (OCTA).
Change From Baseline in branch Neovascularization network in the Study Eye at 2 years | Baseline and 2 years
  The branch neovascularization network in the study eye is evaluated by a central reading center using OCT angiography (OCTA).
Proportion of participants on 12 weeks or more treatment intervals at the end of the study. | End of study (up to 100 weeks)
  Proportions are based on the number of participants who have not discontinued the study at the end of the study. The treatment interval at a given visit is defined as the treatment interval decision followed at that visit.
Number of faricimab injections received from Week 20 until the end of the study. | Week 20 through end of study (up to 100 weeks)
  Count of the number of faricimab injections each participant received after the treatment initiation period (baseline to week 12).
Incidence and severity of ocular adverse events | From first dose of study drug through end of study (up to 104 weeks)
  This analysis of adverse events (AEs) only includes ocular AEs. Investigators sought information on AEs at each contact with the participants. All AEs are recorded and the investigator made an assessment of seriousness, severity, and causality of each AE.
Incidence and severity of Non-Ocular Adverse Event | From first dose of study drug through end of study (up to 104 weeks)
  This analysis of AEs only includes non-ocular (systemic) AEs. Multiple occurrences of the same AE in one individual are counted only once. Investigators sought information on AEs at each contact with the participants. All AEs were recorded and the investigator made an assessment of seriousness, severity, and causality of each AE.

CONTACTS AND LOCATIONS:
Locations (30):
- Italy (7):
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico-Clinica Regina Elena, Milan
  - Medical Retina Service, Operative Unit Ophthalmology - MultiMedica Spa (IRCCSMM), Milan
  - ASST-Fatebenefratelli-Sacco P.O.L. Sacco, Milan
  - Eye Unit, University Hospital Maggiore della Carità, Novara
  - IRCCS Fondazione G.B. Bietti per lo Studio e la Ricerca in Oftalmologia ONLUS,, Roma
  - Department of Ophthalmology, University Vita Salute - Scientific Institute of San Raffaele, San Raffaele
  - Department of Ophthalmology, University of Udine, Udine
- Portugal (10):
  - Espaço Médico de Coimbra, Coimbra
  - Ophthalmology Department, Hospitais Universidade de Coimbra,, Coimbra
  - Unidade Local de Saúde da Região de Leiria, E.P.E., Leiria
  - almPRIMUM- Serviços de Oftalmologia Médica e Cirúrgica, Lisbon
  - Instituto de Retina e Diabetes Ocular de Lisboa (IRL),, Lisbon
  - Serviço de Oftalmologia, Centro Hospitalar Lisboa Norte, Hospital de Santa Maria, Lisbon
  - Unidade Local de Saúde São José, Lisbon
  - ULS-LOD - Hospital Beatriz Ângelo, Loures
  - Department of Ophthalmology, Porto Medical School / Hospital S. João, Porto
  - Serviço Oftalmologia, Centro Hospitalar Universitário de Santo António, E.P.E.,, Porto
- Spain (7):
  - Centro de Oftalmologia Barraquer, Barcelona
  - Hospital Vall d'Hebrón Department of Ophthalmology, Barcelona
  - Institut Català de Retina (ICR), Clinical Trial Unit, Barcelona
  - Valles Ophthalmology Research, S.L., Hospital General de Catalunya,, Barcelona
  - Department of Ophthalmology, Fundación Jiménez Díaz University Hospital, Madrid
  - Instituto Oftalmologico Fernandez-Veja, Oviedo
  - Fundación de Oftalmología Médica de la Comunitat Valenciana (Fom), Valencia
- United Kingdom (6):
  - Clinical Trial Unit, Dep. Ophth., Gloucestershire Hospitals NHS Foundation Trust,, Gloucester
  - Clinical Eye Research Centre - St. Paul's Eye Unit, Royal Liverpool University Hospital, Liverpool
  - Clinical Trial Unit, Dep. Ophth., Gloucestershire Hospitals NHS Foundation Trust, London
  - ICORG - Imperial College Ophthalmologic Research Group, London
  - University Hospital Southampton NHS Foundation Trust, Southampton
  - Wolverhampton and Midland Counties Eye Infirmary, New Cross Hospital, Wolverhampton